CLINICAL TRIAL: NCT04026815
Title: Health Status and Its Socio-economic Covariates of the Older Population in Poland - the Nationwide, Cross-sectional PolSenior2 Survey.
Brief Title: Health Status and Its Socio-economic Covariates of the Older Population in Poland - the Nationwide PolSenior2 Survey.
Acronym: PolSenior2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: Ministry of Health, Poland (Other Government); Medical University of Silesia (Other); Jagiellonian University (Other); International Institute of Molecular and Cell Biology in Warsaw (Unknown); SGH Warsaw School of Economics (Unknown); Medical University of Lodz (Other); National Institute of Public Health-National Institute of Hygiene (Unknown)
Responsible Party: Principal Investigator, Tomasz Zdrojewski, M.D., Ph.D., Assoc. Prof., Medical University of Gdansk
Other Study IDs: 6/5/4.2/NPZ/2017/1203/1257
Record Dates: First submitted 2019-07-15; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Aging Disorder; Age Problem; Healthy Aging; Immunity Disorders; Frailty Syndrome; Behaviors, Health; Health Care Utilization
MeSH Terms: conditions — Immune System Diseases; Frailty; Health Behavior; Patient Acceptance of Health Care | interventions — Health Records, Personal; Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 36 ml of whole blood and 20 ml of urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- 60 - 65 years: Subjects were selected using a three stage stratified and proportional random sampling in seven equally size (n=850) age groups: 60-65, 65-69, 70-74, 75-79, 80-84, 85-89, 90+ years.
  Interventions: Other: medical history, blood and urine tests
- 65 - 69 years: Subjects were selected using a three stage stratified and proportional random sampling in seven equally size (n=850) age groups: 60-65, 65-69, 70-74, 75-79, 80-84, 85-89, 90+ years.
  Interventions: Other: medical history, blood and urine tests
- 70 - 74 years: Subjects were selected using a three stage stratified and proportional random sampling in seven equally size (n=850) age groups: 60-65, 65-69, 70-74, 75-79, 80-84, 85-89, 90+ years.
  Interventions: Other: medical history, blood and urine tests
- 75 - 79 years: Subjects were selected using a three stage stratified and proportional random sampling in seven equally size (n=850) age groups: 60-65, 65-69, 70-74, 75-79, 80-84, 85-89, 90+ years.
  Interventions: Other: medical history, blood and urine tests
- 80 - 84 years: Subjects were selected using a three stage stratified and proportional random sampling in seven equally size (n=850) age groups: 60-65, 65-69, 70-74, 75-79, 80-84, 85-89, 90+ years.
  Interventions: Other: medical history, blood and urine tests
- 85 - 89 years: Subjects were selected using a three stage stratified and proportional random sampling in seven equally size (n=850) age groups: 60-65, 65-69, 70-74, 75-79, 80-84, 85-89, 90+ years.
  Interventions: Other: medical history, blood and urine tests
- ≥90 years: Subjects were selected using a three stage stratified and proportional random sampling in seven equally size (n=850) age groups: 60-65, 65-69, 70-74, 75-79, 80-84, 85-89, 90+ years.
  Interventions: Other: medical history, blood and urine tests

INTERVENTIONS:
Other: medical history, blood and urine tests — The study protocol consists of questionnaires (medical, socio-economic, dietary), comprehensive geriatric assessment, physical examination, anthropometric and blood pressure measurements and laboratory tests.

SUMMARY:
The PolSenior2 survey is aimed to characterise health status of old and very-old adults in Poland.

DETAILED DESCRIPTION:
One of the goals is assessing the prevalence and control of age-related diseases and of the "geriatric giants" (immobility, instability, incontinence, sensory deficiency, cognition and mood disorders) which lead to frailty, disability and dependence. Monitoring of health status, health behaviors and identifying socio-economic factors favoring successful aging will be significant. As the polypragmasy and adverse drug reactions remain a significant issue in the geriatric care, pharmacotherapy and medical adherence will also be examined.

The additional purpose of the study is to evaluate the utilization and access to health care and social services in respect to needs for assistance and long-term care, as well as the level and different forms of these needs.

The project is planned as a cross-sectional survey of representative sample of 6000 people aged 60 years and over. The study protocol consists of questionnaires (medical, socio-economic, dietary), comprehensive geriatric assessment, anthropometric and blood pressure measurements and laboratory tests. The data are collected by well-trained nurses during three visits at respondents homes.

ELIGIBILITY:
Inclusion Criteria:

* over 60 years of age,
* randomly selected from database of all Polish citizens,
* consent to participate in the study.

Exclusion Criteria:

* under 60 years of age,
* no consent to participate in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research population is assumed to include 6000 individuals in seven equivalent age cohorts (60-64 years, 65-69 years, 70-74 years, 75-79 years, 80-84 years, 85-89 years, 90+ years old) with equal representation of males and females in each of them.
  Research participants were randomly recruited in a stratified, proportional draw. The pattern for respondent selection was designed to obtain a population representative for Polish old citizens.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional status as assessed by Vulnerable Elders Survey-13 | baseline
  The Vulnerable Elders Survey-13 (VES-13) is a simple function-based tool for screening community-dwelling populations to identify older persons at risk for health deterioration. The VES-13 considers age, self-related health, limitation in physical function, and functional disabilities. The total possible score ranges from 0 to 10, with higher scores indicating increased disability.
Functional status as assessed by Instrumental Activity of Daily Living | baseline
  This will be assessed using the Instrumental Activity of Daily Living (IADL-Lawton) instrument. IADL evaluates independent living skills. Each activity has specific level of participation that can be selected. Scores range from 0 (low function, dependent) to 8 points (high function, independent).
Functional status as assessed by Activity of Daily Living Index | baseline
  This will be assessed using the Activity of Daily Living (ADL-Katz Index) instrument. ADL evaluates functional status as a measurement of the patient's ability to perform activities of daily living. Each activity is rated as being completed independently or not. Scores range is 0-6 points, higher score is better.
Mood deterioration incidence | baseline
  The Geriatric Depression Scale (GDS) is a 15-item self-report assessment designed specifically to identify symptoms of depression in the elderly. Participants are asked to respond by answering yes or no in reference to how they felt over the past 2 weeks. The score 5 and more suggests the suspicion of depression, higher scores indicate more severe depressive syndrome. The final diagnosis of depression needs clinical assessment.
Cognitive functions as assessed by the Mini Mental State Examination | baseline
  The Mini Mental State Examination (MMSE) investigates specific cognitive functions. Scale range: 0-30. The score 23 and below indicates significant deterioration of cognitive functions and dementia. Score between 24-27 indicates mild cognitive impairment. Normal score ranges between 28-30.
Cognitive functions as assessed by Clock Drawing Test | baseline
  The Clock Drawing Test is a test used for the assessment of cognitive impairment based on sketches of a clock completed by a patient. The assessment is based on identifying abnormalities in the drawings, which may include poor number positioning, omission of numbers, incorrect sequencing, missing clock hands and the presence of irrelevant writing. According to Sunderland the score is: 0-10. Higher score indicates normal cognitive functions.
Comorbidities incidence | baseline
  the prevalence of comorbidities
Nutritional status assessed by the Mini Nutritional Assessment questionnaire (MNA) | baseline
  The MNA is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition. The Screening score(max. 14 points) is 12-14 points indicates "Normal nutritional status", 8-11 points indicates "At risk of malnutrition", 0-7 points indicates "Malnourished". For the full assessment there are proposed scores: 24 pts and more "Normal nutritional status"; 23,5-17 "At risk of malnutrition"; below 17 - malnourished"
Sarkopenia incidence | baseline
  The prevalence of sarcopenia will be assessed by analysis of grip strength (use of dynamometer).

SECONDARY OUTCOMES:
Number of drugs taken | baseline
  assessement of pharmacotherapy and polypragmasy
Medical care availability | five years back from baseline
  number of hospitalizations and of outpatients visits in last five years
Quality of life as assessed by the World Health Organization Quality of Life Age (WHOQOL-AGE) | baseline
  The WHOQOL-AGE has been designed and validated to measure quality of life older adults. It provides a single score that ranges on a 0-100 scale, with higher scores indicating higher quality of life.
Quality and patterns of sleep assessmed by the Pittsburgh Sleep Quality Index | baseline
  The Pittsburgh Sleep Quality Index has been designed and validated to assess the presence of sleep disorders. It includes 19 questions that combine to evaluate 7 components of sleep, each evaluated from 0 to 3 (0 = no difficulty, 3 = severe difficulty). A total score greater than 5 indicates a sleep disorder.
Alcohol abuse assessment | baseline
  Alcohol abuse will be assessed using the Short Michigan Alcohol Screening (SMASM). This 10 item inventory characterizes behavior associated with alcoholism, the higher the score, the greater the severity of alcoholism in a respondent.
Physical activity assessmed by the Seven-Day Recall Physical Activity Questionnaire (PAR) | baseline
  Minutes of physical activity measured by the 7-Day Physical Activity Recall (7-Day PAR), which is an interviewer-administered self-report physical activity measure of minutes spent in moderate and vigorous intensity leisure and non-leisure activities over the preceding 7 days. Low time span (low number of minutes) spent on physical activity suggest low level of it and is one of significant symptoms of frailty syndrome.
Presence and severity of chronic pain assessmed by the Pain Assessment Scale (PAS) | baseline
  measurement by the Pain Assessment Scale (PAS)
Presence and severity of chronic pain assessmed by the Visual Analog Scale (VAS) | baseline
  VAS is a self-assessed maximum pain reported using a 0-100 mm visual analog scale, where 100 signifies maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz R. Zdrojewski, MD, Prof, Principal Investigator — Medical University of Gdansk, Poland
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland